CLINICAL TRIAL: NCT02820402
Title: Project Viva: a Longitudinal Study of Health for the Next Generation
Status: Active, not recruiting | Type: Observational
Sponsor: Harvard Pilgrim Health Care (Other)
Collaborators: Brigham and Women's Hospital (Other); Harvard School of Public Health (HSPH) (Other)
Responsible Party: Sponsor
Other Study IDs: 5R37HD034568 (NIH)
Record Dates: First submitted 2016-03-07; First posted 2016-07-01 (Estimated); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Pediatric Obesity
Keywords: Pregnancy; Obesity; Diet; Maternal/child health; Asthma/allergy; Air pollution; Epigenetics; Cognition/behavior
MeSH Terms: conditions — Pediatric Obesity; Obesity; Asthma; Hypersensitivity; Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Mom: 1st trimester-EDTA top (plasma, RBC, WBC-DNA), heparin top (plasma); 2nd trimester-EDTA top (plasma, RBC, WBC-DNA), heparin top; birth - hair; early childhood-EDTA top (plasma, RBC, WBC-DNA), heparin top (plasma); mid-teen-EDTA top (plasma, RBC, WBC-DNA), heparin top (plasma, RBC), grey top (plasma), urine
  Child: cord blood-heparin top (cell pellets and supernatant), serum, EDTA top (plasma, WBC-DNA); early childhood-EDTA top (plasma, WBC-DNA), heparin top (plasma, RBC); early childhood (Immune Substudy)-EDTA top, heparin top (room temp - stimulation supernatants, plasma), and heparin top (cold - RBC, plasma); mid-childhood-EDTA top (plasma, RBC, WBC-DNA), heparin top (plasma, RBC), grey top (plasma), urine, hair; early teen - EDTA top (plasma, RBC, WBC-DNA), heparin top (plasma, RBC), 2 ml grey top (plasma), urine, hair; mid-teen-EDTA top (plasma, RBC, WBC-DNA), heparin top (plasma, RBC), grey top (plasma), PAXgene blood RNA (RBC), baby teeth, urine, hair
Oversight: Data Monitoring Committee: No

SUMMARY:
Project Viva is a prospective cohort study of maternal and child health, following over 2,000 mother-child pairs from the mother's pregnancy into the child's adolescence.

DETAILED DESCRIPTION:
In 1999-2002 the Project Viva team recruited 2,670 pregnant women during their first trimester of pregnancy from eight obstetric (OB) offices of a multi-site group practice in eastern Massachusetts. 2,128 of the women had a live birth and approximately 1,600 mother-child pairs are still involved in the study. Project Viva collects data annually from multiple sources, including questionnaires, interviews, medical records, examinations, and biospecimen samples. Project Viva intends to follow participants as long as there is grant funding and interest from the participants. Some of the most beneficial health findings come from long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Less than 22 weeks pregnant at the time of enrollment
* Receive prenatal care at one of the selected practices
* Plan on delivering at one of two study hospitals
* Be able to answer questionnaires in English.

Exclusion Criteria:

* Multiple gestation
* Plans to move away before delivery
* Plans to terminate the pregnancy

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Mothers initially recruited during their first prenatal visit (median 9.9 wks gestation) at a multi-specialty group practice in eastern Massachusetts between 1999-2002 and their children.
  Project Viva recruited 2670 women (64% of those who were approached for participation). 2,128 were still enrolled at the time of delivery and had live births, resulting in a cohort of 2,128 mother-child pairs.
Sampling Method: Non-Probability Sample
Enrollment: 2128 (Actual)
Dates: Start 1999-01 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Cross-sectional and longitudinal measurements of child BMI z-score in kg/m^2, standardized into a sex- and age-specific z-score using national reference data (CDC growth charts) | Research measurements at birth, 6mo, early childhood (~3y), mid-childhood (~8y), early teen (~14y), and mid-late teen (~17y).
  The study team measures child weight and length/height at each time point, and BMI is calculated and standardized based on the child's age at the time of measurement.
Maternal post-partum weight retention, calculated as the difference between weight in kg at 1 year postpartum and pre-pregnancy weight | Before the Project Viva pregnancy and 1-year postpartum
  Investigators obtained prenatal weights from the clinical record, and calculated total gestational weight gain (GWG) as the difference between the last weight recorded in the 4 weeks prior to delivery and pre-pregnancy weight. Project Viva mothers reported their weight at 1-year postpartum via questionnaire.
Child metabolic risk score, calculated as a standard deviation (SD) score | HDL-cholesterol, triglycerides, insulin, glucose and waist circumference measured at ~8y, ~14y, and ~17y of age. Blood pressure measured at birth, ~6mo, ~3y, ~8y, ~14y, and ~17y. Metabolic risk score calculated at ~8y, ~14y, and ~17y.
  Investigators derived the metabolic risk score as the mean of 5 sex- and cohort-specific z-scores for: waist circumference (cm), systolic blood pressure (SBP, calculated as the average of 5 measurements taken 1 minute apart), HDL cholesterol (mg/dL, scaled inversely), log-transformed triglycerides (mg/dL) and log-transformed HOMA-IR (calculated as fasting insulin [μU/mL] x fasting glucose [mg/dL]/405).
Child neurodevelopment, assessed by continuous scores on the Wide Range Assessment of Memory and Learning, Second Edition (WRAML2), Design and Picture Memory subtests and The Kaufman Brief Intelligence Test, Second Edition (KBIT-2) | Children completed both the WRAML2 and the KBIT-2 at the mid-childhood visit (~8y)
Mother's report of a clinical diagnosis of asthma, wheeze or reactive airway disease | Interviews administered at 6mo, early childhood (~3y), mid-childhood (~8y), early teen (~14y), and mid-late teen (~17y).
  Mothers answered yes or no when asked "have you ever been told by a health care professional, such as a doctor, physician assistant or nurse practitioner, that your child has…
  1. Asthma?
  2. Wheezing or reactive airways?
  Mothers reported asthma, wheezing and reactive airways as a single outcome at the infancy visit and separately at the early and mid-childhood visits. At the early teen visit, the mother reported a diagnosis of asthma only.

SECONDARY OUTCOMES:
Child's birth length in cm | Measured at birth
Child's birth weight in grams, standardized into a sex- and gestational age-specific z-score using national reference data | Measured at birth

CONTACTS AND LOCATIONS:
Overall Officials: Emily Oken, MD, MPH, Principal Investigator — Harvard Medical School / Harvard Pilgrim Health Care Institute

IPD SHARING:
Plan to Share IPD: Yes
Project Viva protocols include a data sharing plan. The process for requesting data is detailed in the study policy document, available on the Project Viva website: https://www.hms.harvard.edu/viva/policies-for-using-our-data.pdf.

REFERENCES:
- [Derived] Harnois-Leblanc S, Rifas-Shiman SL, Switkowski KM, Perng W, Aris IM, Oken E, Young JG, Hivert MF. Estimating sex-specific population-level effects of limiting sugar-sweetened beverages or 100% fruit juices during childhood on insulin resistance, central adiposity, and glycemic outcomes in late adolescence. Am J Epidemiol. 2025 Oct 18:kwaf225. doi: 10.1093/aje/kwaf225. Online ahead of print. PMID 41108089
- [Derived] Switkowski KM, Kronsteiner-Gicevic S, Rifas-Shiman SL, Lightdale JR, Oken E. Evaluation of the Prime Diet Quality Score from Early Childhood Through Mid-Adolescence. J Nutr. 2024 Jun;154(6):1890-1906. doi: 10.1016/j.tjnut.2024.04.014. Epub 2024 Apr 16. PMID 38614240
- [Derived] Choudhary D, Rideout TC, Cameron CE, Lehman HK, Oken E, Rifas-Shiman SL, Wen X. Egg Introduction during Infancy is Associated with Lower Fat Mass Index in Females at Early Adolescence. J Nutr. 2023 Jan;153(1):158-166. doi: 10.1016/j.tjnut.2022.11.003. Epub 2022 Dec 20. PMID 36913449
- [Derived] McGovern C, Rifas-Shiman SL, Switkowski KM, Woo Baidal JA, Lightdale JR, Hivert MF, Oken E, Aris IM. Association of cow's milk intake in early childhood with adiposity and cardiometabolic risk in early adolescence. Am J Clin Nutr. 2022 Aug 4;116(2):561-571. doi: 10.1093/ajcn/nqac103. PMID 35441227
- [Derived] Wu AJ, Aris IM, Rifas-Shiman SL, Oken E, Taveras EM, Hivert MF. Longitudinal associations of fruit juice intake in infancy with DXA-measured abdominal adiposity in mid-childhood and early adolescence. Am J Clin Nutr. 2021 Jul 1;114(1):117-123. doi: 10.1093/ajcn/nqab043. PMID 33829237
- [Derived] Switkowski KM, Camargo CA, Rifas-Shiman SL, Fuller H, Oken E. Early-Life Factors Are Associated with Vitamin D Status in Early and Mid-Childhood and May Differ between White and Black Children. J Nutr. 2021 May 11;151(5):1256-1268. doi: 10.1093/jn/nxaa456. PMID 33693813
- [Derived] Turturice BA, Theorell J, Koenig MD, Tussing-Humphreys L, Gold DR, Litonjua AA, Oken E, Rifas-Shiman SL, Perkins DL, Finn PW. Perinatal granulopoiesis and risk of pediatric asthma. Elife. 2021 Feb 10;10:e63745. doi: 10.7554/eLife.63745. PMID 33565964
- [Derived] Mahmassani HA, Switkowski KM, Scott TM, Johnson EJ, Rifas-Shiman SL, Oken E, Jacques PF. Maternal Intake of Lutein and Zeaxanthin during Pregnancy Is Positively Associated with Offspring Verbal Intelligence and Behavior Regulation in Mid-Childhood in the Project Viva Cohort. J Nutr. 2021 Mar 11;151(3):615-627. doi: 10.1093/jn/nxaa348. PMID 33484136
- [Derived] Gingras V, Aris IM, Rifas-Shiman SL, Switkowski KM, Oken E, Hivert MF. Timing of Complementary Feeding Introduction and Adiposity Throughout Childhood. Pediatrics. 2019 Dec;144(6):e20191320. doi: 10.1542/peds.2019-1320. PMID 31757860
- [Derived] Switkowski KM, Jacques PF, Must A, Fleisch A, Oken E. Associations of protein intake in early childhood with body composition, height, and insulin-like growth factor I in mid-childhood and early adolescence. Am J Clin Nutr. 2019 Apr 1;109(4):1154-1163. doi: 10.1093/ajcn/nqy354. PMID 30869114
- [Derived] Gingras V, Rifas-Shiman SL, Taveras EM, Oken E, Hivert MF. Dietary behaviors throughout childhood are associated with adiposity and estimated insulin resistance in early adolescence: a longitudinal study. Int J Behav Nutr Phys Act. 2018 Dec 17;15(1):129. doi: 10.1186/s12966-018-0759-0. PMID 30558613
- [Derived] Gingras V, Rifas-Shiman SL, Derks IPM, Aris IM, Oken E, Hivert MF. Associations of Gestational Glucose Tolerance With Offspring Body Composition and Estimated Insulin Resistance in Early Adolescence. Diabetes Care. 2018 Dec;41(12):e164-e166. doi: 10.2337/dc18-1490. Epub 2018 Oct 16. No abstract available. PMID 30327360
- [Derived] Switkowski KM, Jacques PF, Must A, Hivert MF, Fleisch A, Gillman MW, Rifas-Shiman S, Oken E. Higher Maternal Protein Intake during Pregnancy Is Associated with Lower Cord Blood Concentrations of Insulin-like Growth Factor (IGF)-II, IGF Binding Protein 3, and Insulin, but Not IGF-I, in a Cohort of Women with High Protein Intake. J Nutr. 2017 Jul;147(7):1392-1400. doi: 10.3945/jn.117.250589. Epub 2017 Jun 7. PMID 28592512
- [Derived] Switkowski KM, Jacques PF, Must A, Kleinman KP, Gillman MW, Oken E. Maternal protein intake during pregnancy and linear growth in the offspring. Am J Clin Nutr. 2016 Oct;104(4):1128-1136. doi: 10.3945/ajcn.115.128421. Epub 2016 Aug 31. PMID 27581477
- See also: Full publication list from Project Viva website — https://www.hms.harvard.edu/viva/project-viva-publication-list.html